CLINICAL TRIAL: NCT02726867
Title: Evaluation of Efficacy and Safety of Levetiracetam, Lacosamide and Ketamine as Adjunctive Treatment of Refractory Status Epilepticus
Brief Title: Levetiracetam, Lacosamide and Ketamine as Adjunctive Treatment of Refractory Status Epilepticus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Responsible Party: Principal Investigator, Pavel Klein, M.D., Mid-Atlantic Epilepsy and Sleep Center, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAES-003
Record Dates: First submitted 2014-12-12; First posted 2016-04-04 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy; Status Epilepticus
Keywords: refractory status epilepticus; levetiracetam; lacosamide; ketamine
MeSH Terms: conditions — Epilepsy; Status Epilepticus | interventions — Levetiracetam; Lacosamide; Ketamine; Phenobarbital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- levetiracetam (Active Comparator): Patients with status epilepticus who have been treated with standard dose lorazepam (or midazolam) and ≥ 1000 mg phenytoin with documented levels of ≥20 mg/ml and continue to have clinical SE for ≥1-24 hours after phenytoin loading will receive intravenously (i.v.) 4000 mg levetiracetam.
  Interventions: Drug: levetiracetam
- lacosamide (Active Comparator): Patients with status epilepticus who have been treated with standard dose lorazepam (or midazolam) and ≥ 1000 mg phenytoin with documented levels of ≥20 mg/ml and continue to have clinical SE for ≥1-24 hours after phenytoin loading will receive intravenously (i.v.) 600 mg lacosamide.
  Interventions: Drug: lacosamide
- ketamine (Active Comparator): Patients with status epilepticus who have been treated with standard dose lorazepam (or midazolam) and ≥ 1000 mg phenytoin with documented levels of ≥20 mg/ml and continue to have clinical SE for ≥1-24 hours after phenytoin loading will receive intravenously (i.v.) 2.5 mg/kg ketamine.
  Interventions: Drug: Ketamine
- phenobarbital (Active Comparator): Patients with status epilepticus who have been treated with standard dose lorazepam (or midazolam) and ≥ 1000 mg phenytoin (PHT) with documented levels of ≥20 mg/ml and continue to have clinical SE for ≥1-24 hours after PHT loading will receive intravenously (i.v.) phenobarbital 15 mg/kg.
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: levetiracetam — Treatment will consist of LEV 4000 mg i.v. over 10 minutes.
  Other Names: Keppra
  Arms: levetiracetam
Drug: lacosamide — Treatment will consist of LCM 600 mg i.v. over 10 minutes
  Other Names: Vimpat
  Arms: lacosamide
Drug: Ketamine — Treatment will consist of KET 2.5 mg/kg over 10 minutes
  Other Names: Ketalar
  Arms: ketamine
Drug: Phenobarbital — Treatment will consist of PHB 15 mg/kg mg i.v. at 100 mg/minute rate
  Other Names: Phenobarb
  Arms: phenobarbital

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of levetiracetam , lacosamide and ketamine treatment of refractory status epilepticus. This will be a randomized, open-label, four-arm pilot study comparing time to cessation of refractory status epilepticus, determined by continuous EEG monitoring, in patients with refractory status epilepticus. Patients with status epilepticus who have been treated with standard dose lorazepam (or midazolam) and ≥ 1000 mg phenytoin with documented levels of ≥20 mg/ml and continue to have clinical status epilepticus for ≥1-24 hours after phenytoin loading will receive intravenously (i.v.) either 4000 mg levetiracetam, 600 mg lacosamide (Group B), 2.5 mg/kg ketamine or phenobarbital 15 mg/kg phenobarbital (Group D)

DETAILED DESCRIPTION:
40 18-70 year old men and women with refractory status epilepticus, defined as status epilepticus continuing for >1 hour after completion of standard treatment with lorazepam (or midazolam) and i.v. phenytoin (or fos-phenytoin),will be enrolled. Participants will be randomized into four treatment arms, levetiracetam 4000 (Group A, n=10), lacosamide 600 mg (Group B, n=10), ketamine 2.5 mg/kg (group C,n=10),and phenobarbital 15 mg/kg (Group D, n=10) in a 1:1:1:1 ratio. Baseline evaluations will include continuous EEG, phenytoin levels prior to study intervention, CBC, CMP, serum Ca, Po4 and Mg.

Treatment will consist of levetiracetam 4000 mg i.v. over 10 minutes, lacosamide 600 mg i.v. over 10 minutes, ketamine 2.5 mg/kg over 10 minutes, or phenobarbital 15 mg/kg mg i.v. at 100 mg/minute rate.

Participants will be evaluated with ongoing physical examination and continuous EEG monitoring. Continuous EEG monitoring will be started before initiation of the study treatment, with documentation of electrographic status epilepticus. It will continue throughout the treatment period. Subjects will be observed for 1 hour clinically and with continuous EEG monitoring for cessation of SE. Participants in whom status epilepticus stops within 60 minutes of completion of study treatment will continue to receive phenytoin (150 mg i.v. q 12 hours, standard dose) and the study medication (levetiracetam 1500 mg i.v. q 12 hourly, lacosamide 300 mg q 12 hourly, ketamine 50 mg qid (vs. 40 mcg/kg/min i.v. infusion, as clinically applicable, or phenobarbital 90 mg i.v. q 12 hourly). Continuous EEG monitoring will continue for 72 hours to monitor for relapse of status epilepticus. Participants in whom status epilepticus fails to stop within 60 minutes after completion of study treatment ("non-responders") will undergo standard treatment with medically-induced coma, with intubation/ventilation and i.v. midazolam or propofol treatment at a dose to be titrated to EEG effect of "burst suppression" or suppression of all background activity. All patients, responders and non-responders alike, will continue treatment with phenytoin i.v., 150 mg q 12 hourly or, for conscious patients, 300 mg p.o. qhs for 72 hours after completion of study treatment. In patients requiring medical coma after study treatments (non-responders), medical coma will be discontinued after 48 hours. All participants will continue to be monitored with continuous EEG for 72 hours from completion of study treatment. If status epilepticus returns during this time, medical coma will be re-instituted and patients will be treated according to standard clinical care for prolonged SE

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Ability and willingness by surrogates to signed informed consent form.
3. Clinically and electrographically documented ongoing SE lasting ≥1 hour- ≤24 hours

Exclusion Criteria:

1. Creatinine > 2.5 mg/dl
2. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, metabolic or endocrine disturbances, renal or liver disease
3. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements
4. Pregnancy
5. Inability or unwillingness of subject or legal surrogate to give written informed consent
6. Known allergy to a study drug
7. Hypo- or hyperglycemia as cause of SE

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cessation of status epilepticus by EEG. | 60 minutes
  The cessation of ictal epileptic EEG activity measured by EEG.

SECONDARY OUTCOMES:
Cessation of status epilepticus by clinical examination | 60 minutes
  Measurement of the time to status epilepticus cessation by clinical examination.

OTHER OUTCOMES:
Recurrence of status epilepticus. | 72 hours
  The recurrence of status epilepticus in responders in during the 72 hours of monitoring.
Rate of early treatment discontinuation | 72 hours
  Rate of treatment discontinuation within 72 hours.
Duration of hospitalization | 3 months
  Investigators will count the number days of hospitalization.
Number of participants with neurological deficit. | 3 months
  Investigators will identify the number of patients with neurological deficit at 3 months are the other measure outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.D., Principal Investigator — Mid-Atlantic Epilepsy and Sleep Center
Locations (1):
- MidAtlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States